CLINICAL TRIAL: NCT07199192
Title: A Multicenter, Randomized, Controlled Trial to Evaluate the Effectiveness and Safety of Systemic Corticosteroid Treatment for Hospitalized Patients With Severe Acute Respiratory Infection and Hypoxemia (STRIVE 003)
Brief Title: Steroid Treatment for Severe Acute Respiratory Infection (STAR) Trial
Acronym: STAR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STRIVE 003
Record Dates: First submitted 2025-09-17; First posted 2025-09-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hypoxemia; Severe Acute Respiratory Syndrome
MeSH Terms: conditions — Hypoxia; Severe Acute Respiratory Syndrome | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corticosteroid Group (Experimental): Participants in the corticosteroid group will receive systemic corticosteroids at a dose equivalent to 40 mg of prednisolone per day for 7 days or until discharge, whichever is sooner. Clinicians will select the systemic corticosteroid medication and the route of administration.
  Interventions: Drug: Corticosteroid
- Control Group (No Intervention): Participants in the no corticosteroid group will not receive systemic corticosteroids for 7 days or until hospital discharge, whichever is sooner, unless (i) they meet prespecified criteria for the administration of systemic corticosteroids (e.g., anaphylaxis) or (ii) their clinicians determine that the administration of systemic corticosteroids is required for the optimal care of the participant for other reasons.

INTERVENTIONS:
Drug: Corticosteroid — systemic corticosteroids at a dose equivalent to 40 mg of prednisolone per day for 7 days or until discharge
  Arms: Corticosteroid Group

SUMMARY:
Multicenter, parallel-group, randomized clinical trial comparing the administration of systemic corticosteroids at a dose equivalent to 40 mg of prednisolone per day for 7 days vs no corticosteroid administration among adults hospitalized with severe acute respiratory infection and hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Severe acute respiratory infection (SARI), defined as a suspected infection of the respiratory tract that meets each of the following 4 criteria:

  1. Onset in the last 10 days AND
  2. Results in hospitalization AND
  3. At least one symptom or sign of respiratory illness (defined as purulent sputum, new or worsened cough, new or worsened dyspnea, tachypnea with respiratory rate ≥22 breaths per minute, rales, or bronchial breath sounds) AND
  4. At least one symptom or sign of acute infection (defined as a temperature ≥38°C or ≤36°C, feverishness, chills, altered mental status, a white blood cell count of >12,000/mm3, <4,000/mm3, or >10% immature neutrophils, or imaging findings consistent with acute respiratory infection).
* Hypoxemia, defined as meeting one or more of the following at the time of eligibility assessment:

  1. An oxygen saturation <92% in a patient who does not receive chronic supplemental oxygen OR
  2. Receipt of ≥3 liters per minute of supplemental oxygen or a fraction of inspired oxygen of ≥0.35 in a patient who does not receive chronic supplemental oxygen OR
  3. Receipt of a flow rate of supplemental oxygen ≥3 liters per minute greater than pre-illness baseline or a fraction of inspired oxygen ≥0.10 greater than pre-illness baseline in a patient who receives chronic supplemental oxygen.

Exclusion Criteria:

* Hospitalized for >72 hours
* Primary etiology of hypoxemia is a condition other than respiratory infection
* Known allergy or adverse reaction to systemic corticosteroids
* Known active infection with SARS-CoV-2, known active infection with Pneumocystis jirovecii, or another established indication for systemic corticosteroids
* Known active disseminated or pulmonary infection with Mycobacterium tuberculosis, Aspergillus, Blastomyces, Coccidioides, Cryptococcus, Histoplasma, or Strongyloides species; active systemic infection with herpes simplex virus, varicella zoster virus, or cytomegalovirus; or another established contraindication to systemic corticosteroids
* Prisoner
* Treatment is prioritizing end-of-life symptom management over prolongation of life
* Investigator determines that participation in the trial is not in the patient's best interest
* Receipt of greater than 14 days of systemic corticosteroids at a dose equivalent to greater than 10 mg of prednisolone per day in the 30 days prior to hospital presentation (i.e., chronic corticosteroids)
* Receipt of systemic corticosteroids at a dose equivalent to greater than 30 mg of prednisolone per day on 2 or more calendar days since hospital presentation
* Clinicians determine that the administration of systemic corticosteroids at a dose equivalent to greater than 10 mg of prednisolone per day is required, or is likely to be required in the next 24 hours, for the optimal care of the patient (such as for acute exacerbation of chronic obstructive pulmonary disease, adrenal insufficiency, asthma, continuation of chronic corticosteroid therapy, or severe shock)
* Clinicians determine that the administration of systemic corticosteroids is not consistent with the optimal care of the patient (such as for recent peptic ulcer disease, recent gastrointestinal bleeding, severe burns, severe delirium, severe hyperglycemia or diabetic ketoacidosis, or severe hypertension)
* Patient (or surrogate decision-maker / legally authorized representative) declines to provide informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
28-day in-hospital mortality | Day 28
  defined as death from any cause between randomization (Day 0) and 28 days (the end of Study Day 27. Outcome ascertainment ends at hospital discharge.
Advanced respiratory support | Day 28
  receipt of extracorporeal membrane oxygenation (ECMO), IMV, noninvasive mechanical ventilation, or high-flow nasal cannula (HFNC) at a rate of ≥30 liters per minute and a fraction of inspired oxygen of ≥0.4. Mechanical ventilation received solely to facilitate the performance of a procedure (e.g., mechanical ventilation for general endotracheal anesthesia limited to the performance of a surgery) will not qualify. Noninvasive mechanical ventilation received solely for the treatment of obstructive sleep apnea or obesity hypoventilation syndrome will not qualify.
Duration of advanced respiratory support | Day 28
  calculated as a count of calendar days, beginning with the Study Day on which the participant first received advanced respiratory support and ending with the Study Day on which the participant last received advanced respiratory support during the outcome window. Outcome ascertainment ends at hospital discharge.
Duration of hospitalization | Day 28
  calculated as the number of calendar days on which the participant is physically located in a short-term acute care hospital beginning at the time of randomization (Day 0) and ending with the Study Day on which the participant was discharged from the hospital during the outcome window

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Semler, MD, Principal Investigator — Vanderbilt University Medical Center; Jane O'Halloran, MD, PhD, Principal Investigator — Washington Univeristy School of Medicine (ID-CRU)
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No